CLINICAL TRIAL: NCT01442220
Title: Genome-wide Association Study of Pituitary Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, Doctor, Huashan Hospital
Other Study IDs: KY2011-277
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Pituitary Adenomas
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pituitary adenomas is a very common disease, but the cause and genetics hasn't been identified. The investigators are going to use genome-wide association study to identify genes that may be related to pituitary adenomas.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with pituitary adenomas

Exclusion Criteria:

* patients with a family history of endocrine tumors

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with pituitary adenomas and healthy controls will be included.
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-06 (Estimated); Study Completion 2014-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhao, M.D., Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China